CLINICAL TRIAL: NCT05218486
Title: Evaluation of The Effect of Oral Isotretinoin on The Level of Serum YKL40 in Acne Vulgaris Patients
Brief Title: Effect of Oral Isotretinoin on The Level of SerumYKL40 in Acne Vulgaris Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alshimaa Abbas Mohamed Ebrahim (Other)
Responsible Party: Sponsor-Investigator, Alshimaa Abbas Mohamed Ebrahim, principal investigator, Aswan University
Organization: Aswan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 551/7/21
Record Dates: First submitted 2022-01-05; First posted 2022-02-01 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isotretinoin group (Active Comparator): Patients will be treated with Isotretinoin in a dose (from 20 to 40) for 3 months and serum YKL40 will be assessed before and after treatment
  Interventions: Drug: Isotretinoin
- Control group (No Intervention): Assessment of serum YKL40 in healthy individuals

INTERVENTIONS:
Drug: Isotretinoin — Isotretinoin is a vitamin-A derivative for treatment of moderate to severe acne used in a dose from 20-40 mg for 3 months duration
  Arms: Isotretinoin group

SUMMARY:
The aim of the study is to evaluate the effect of oral isotretinoin on SerumYKL40 in acne vulgaris patients.

DETAILED DESCRIPTION:
Acne vulgaris is a common chronic inflammatory disease of the skin. It is found in about 80% of young adults and adolescents. It is a disease that affects the pilosebaceous units of the skin and may result in inflammatory or non-inflammatory lesions,Oral isotretinoin (13-cis-retinoic acid) is the only drug that counteracts all the pathogenetic mechanisms that contribute to the development of acne .The standard dose of isotretinoin is 0.5 to 1 mg/kg per day for 4 months to a cumulative dose of 120-140 mg/kg is effective in the management of acne vulgaris The scope of our study is to detect serum YKL-40 level in acne patient before and after oral isotretinoin treatment

ELIGIBILITY:
Inclusion Criteria:

1. Healthy persons of both sexes with moderate and severe acne.
2. Age above 14 years.

Exclusion Criteria:

1. Pregnant and lactating women, immunocompromised patients.
2. History of chronic liver disease, hyperlipidemia, non-inflammatory acne conditions, , history of neurologic disorders, history of neoplastic disorders, and history of cardiac disease.
3. History of systemic acne treatment for at least 4 weeks prior to inclusion and no topical treatments for at least 2 weeks.
4. Cases with known hypersensitivity reaction to isotretinoin.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effect of oral isotretinoin on SerumYKL40 in acne vulgaris patients. | 3 months
  Assessment in serum level YKL40 level in acne vulgaris patients after isotretinoin therapy with assesment of its level before starting therapy for detecting changes in serum YKL40 and effect of isotretinoin therapy on it.

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan university, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No